CLINICAL TRIAL: NCT02915159
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Subcutaneous Abatacept in Adults With Active Primary Sjögrens Syndrome
Brief Title: A Study to Assess the Efficacy and Safety of Abatacept in Adults With Active Primary Sjögrens Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM101-603; 2016-001948-19 (EudraCT Number)
Record Dates: First submitted 2016-09-23; First posted 2016-09-26 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-07

CONDITIONS: Sjogrens Disease
MeSH Terms: interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abatacept (Experimental): Abatacept for subcutaneous injection 125mg/mL in 1 mL pre-filled syringe for 6 months followed by Open-Label Abatacept for subcutaneous injection 125mg/mL in 1 mL pre-filled syringe for 6 months
  Interventions: Biological: Abatacept
- Placebo (Placebo Comparator): Placebo for Abatacept for subcutaneous injection 125mg/mL in 1 mL pre-filled syringe for 6 months followed by Open-Label Abatacept for subcutaneous injection 125mg/mL in 1 mL pre-filled syringe for 6 months
  Interventions: Biological: Abatacept; Other: Placebo

INTERVENTIONS:
Biological: Abatacept
  Other Names: Orencia; Bristol-Myers Squibb (BMS)-188667
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of abatacept compared to placebo in patients with Sjögren's Syndrome.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) score of at least 5
* Positive anti-SS-A/Ro antibody at screening
* meet the 2016 American College of Rheumatology (ACR) / European League Against Rheumatism Classification Criteria for Sjögren's Syndrome (EULAR SS)

Exclusion Criteria:

* Secondary Sjögrens syndrome
* Active life-threatening or organ-threatening complications of Sjögren's-syndrome
* Other medical condition associated with sicca syndrome

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2019-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (70):
- United States (19):
  - St. Jude Hospital Yorba Linda, Fullerton, California
  - Riverside Medical Clinic, Riverside, California
  - Colorado Arthritis Associates, Lakewood, Colorado
  - North Georgia Rheumatology Group, Lawrenceville, Georgia
  - Intermountain Research Center Inc., Boise, Idaho
  - Johns Hopkins University, Baltimore, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - St. Paul Rheumatology, P.A., Eagan, Minnesota
  - Northwell Health, Great Neck, New York
  - Local Institution, Charlotte, North Carolina
  - Joint and Muscle Medical Care and Research Institute (JMMCRI), Charlotte, North Carolina
  - Duke Clinical Research Unit, Duke Univ Med Ctr, Duke South, Durham, North Carolina
  - Health Research Of Oklahoma, Oklahoma City, Oklahoma
  - East Penn Rheumatology, Bethlehem, Pennsylvania
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - West Tennessee Research Institute, Jackson, Tennessee
  - Metroplex Clinical Research Center, Dallas, Texas
  - Scott Zashin Inc., Dallas, Texas
- Argentina (6):
  - Organizacion Medica De Investigacion S.A. (Omi), Capital Federal, Buenos Aires
  - Local Institution, Ciudad Autonoma Beunos Aires, Buenos Aires
  - Instituto de Asistencia Reumatologica Integral, San Fernando, Buenos Aires
  - Local Institution, Buenos Aires
  - Consultorios Medicos Dr. Catalan Pellet, CABA
  - Instituto Reumatologico Strusberg, Córdoba
- Australia (4):
  - Local Institution, Maroochydore, Queensland
  - Local Institution, Woodville, South Australia
  - Local Institution, Camberwell, Victoria
  - Local Institution, Nedlands, Western Australia
- Brazil (4):
  - Local Institution, Vitória, Espírito Santo
  - Local Institution, Savaldor, Estado de Bahia
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, São Paulo
- Revmatologie s.r.o., Brno, Czechia
- France (7):
  - Local Institution, Bordeaux
  - Local Institution, Le Kremlin-Bicêtre
  - Hopital Europeen, Marseille
  - Local Institution, Marseille
  - Hopital Lapeyronie, Montpellier
  - Local Institution, Paris
  - Local Institution, Strasbourg
- Germany (3):
  - Medizinische Universitaetsklinik Freiburg, Freiburg im Breisgau
  - Med Hochschule Hannover, Hanover
  - Krankenhaus St. Josef, Wuppertal
- Italy (2):
  - Local Institution, Milan
  - Ospedale Santa Maria Della Misericordia, Udine
- Japan (14):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Kitakyushu-shi, Fukuoka
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Nishinomiya-shi, Hyōgo
  - Local Institution, Tsukuba, Ibaraki
  - Local Institution, Kamigyō-ku, Kyoto
  - Local Institution, Sendai, Miyagi
  - Local Institution, Nagasaki, Nagasaki
  - Local Institution, Kurashiki-shi, Okayama-ken
  - Local Institution, Hamamatsu, Shizuoka
  - Local Institution, Chuo-ku, Tokyo
  - Local Institution, Itabashi-ku, Tokyo
  - Local Institution, Meguro-ku, Tokyo
  - Local Institution, Shinjuku-Ku, Tokyo
- Mexico (4):
  - Consultorio Medico de Reumatologia Dr.Jesus Alberto Lopez Garcia, León, Guanajuato
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Local Institution, Distrito Federal
  - Centro de Alta Especialidad en Reumatologia e Investigacion del Potosi S.C., San Luis Potosí City
- Local Institution, San Juan, Puerto Rico
- South Korea (3):
  - Local Institution, Daegu
  - Local Institution, Gwangju
  - Local Institution, Seoul
- Sweden (2):
  - Local Institution, Solna
  - Local Institution, Uppsala

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 250 enrolled; 188 Randomized, 62 not Randomized:Reasons Not randomized: 6 withdrew consent, 1 lost to follow-up, 49 no longer meet study criteria, 6 screening failures
Groups:
- Abatacept - Double Blind Treatment Period: Double Blind Treatment Period SC injection 125mg/mL in 1 mL pre-filled syringe
- Placebo - Double Blind Treatment Period: Double Blind Treatment Period SC injection in 1 mL pre-filled syringe
Period: Overall Study
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Started | 92 | 95
Completed | 81 | 87
Not Completed | 11 | 8
Not completed — Participant no longer meets criteria | 2 | 0
Not completed — poor/non-compliance | 1 | 0
Not completed — Participant withdrew consent | 5 | 1
Not completed — Request to discontinue treatment | 1 | 2
Not completed — Adverse Event | 2 | 2
Not completed — Lack of Efficacy | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period | Total
Number analyzed (Participants) | 92 | 95 | 187
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.2 (12.3) | 52.9 (13.5) | 52.0 (12.9)
Age, Customized [Count of Participants; unit: Participants] — Categorical Age Dispersion Population: Total Participants will = 187 total participants, when the two values assessing the variation in the 65 years group are summed up as well as the two values assessing the variation in the 50 years group are summed up.
  Participants
    < 65 years | 80 | 73 | 153
    ≥ 65 years | 12 | 22 | 34
    ≤ 50 years | 42 | 42 | 84
    > 50 years | 50 | 53 | 103
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 92 | 177
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 10 | 13 | 23
  Unknown or Not Reported | 80 | 77 | 157
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 21 | 23 | 44
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 9 | 19
  White | 60 | 60 | 120
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI)
Description: The EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) total score is calculated as the sum of scores for activity level for each domain.
  The EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) Scoring Algorithm.
  Domain: (Score) Constitutional: (No=0, Low=3, Moderate=6) Lymphadenopathy: (No=0, Low=4, Moderate=8, High=12) Glandular: (No=0, Low=2, Moderate=4) Articular: (No=0, Low=2, Moderate=4, High=6) Cutaneous: (No=0, Low=3, Moderate=6, High=9) Pulmonary: (No=0, Low=5, Moderate=10, High=15) Renal: (No=0, Low=5, Moderate=10, High=15) Muscular: (No=0, Low=6, Moderate=12, High=18) Peripheral Nervous System (PNS): (No=0, Low=5, Moderate=10, High=15) Central Nervous System (CNS): (No=0, Moderate=10, High=15) Haematological: (No=0, Low=2, Moderate=4, High=6) Biological: (No=0, Low=1, Moderate=2)
  (No = No Disease Activity (DA), Low = Low DA, Moderate = Moderate DA, High = High DA)
  Overall score, which can range from 0 to 123, a higher score indicates more disease activity
Time Frame: Day 169
Population: Modified Intent-to-treat (ITT) analysis population: all randomized participants who receive at least one dose of study medication.
Measure: Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
Score on a Scale | -3.2 [-4.6 to -1.9] | -3.7 [-5.0 to -2.4]
Statistical Analysis 1: Comparison: Abatacept - Double Blind Treatment Period vs Placebo - Double Blind Treatment Period; Test type: Superiority; p = 0.4421, longitudinal repeated measures analysis

2. Secondary Outcome: Change From Baseline in EULAR Sjogren's Syndrome Patient Reported Inde (ESSPRI)
Description: The total score EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI) is calculated as the mean of the 3 individual components.
  Total Score Range (0 = Best outcome and 10 = Worst Outcome)
  The scores for the ESSPRI individual components will be used as such reported by the participants and entered in the case report form (CRF), without any further calculations. It consists of 3 questions covering cardinal symptoms of Sjögren's syndrome: dryness, fatigue and pain. Each domain scored on scale of 0-10 (0 =no symptom at all and 10 = worst symptom imaginable), and overall score is calculated as the mean of 3 individual domains.
Time Frame: Day 169
Population: Modified ITT Population
Measure: Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
Score on a Scale | -1.26 [-1.88 to -0.64] | -1.52 [-2.12 to -0.93]
Statistical Analysis 1: Comparison: Abatacept - Double Blind Treatment Period vs Placebo - Double Blind Treatment Period; Test type: Superiority; p = 0.3367, longitudinal repeated measures analysis

3. Secondary Outcome: Change From Baseline in the Stimulated Whole Salivary Flow
Description: The mean change from baseline in the stimulated whole salivary flow at Day 169
Time Frame: Day 169
Population: Modified ITT Population with Stimulated Whole Salivary Flow of at Least 0.1 mL/min at Both Screening and Baseline
Measure: Mean (95% Confidence Interval); unit: mL/min
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 88 | 88
mL/min | 0.057 [-0.115 to 0.230] | 0.108 [-0.060 to 0.276]
Statistical Analysis 1: Comparison: Abatacept - Double Blind Treatment Period vs Placebo - Double Blind Treatment Period; Test type: Superiority; p = .5841, longitudinal repeated measures analysis

4. Secondary Outcome: Change From Baseline of DAS28-C-reactive Peptide (CRP): In The Full Population
Description: The disease activity score DAS28-CRP is a continuous variable which is a composite of 4 variables: the 28 tender joint count (tender28), the 28 swollen joint count (swollen28), CRP and participant assessment of disease activity measure on a visual analogue scale (VAS) of 100mm.
  DAS28-CRP = 0.56 * sqrt(tender28) + 0.28 * sqrt(swollen28) + 0.36 * ln(hsCRP+1) + 0.014 * VAS + 0.96.
  (sqrt = Square root, ln = natural log)
  Positive Scores = Increased Disease Activity Negative Scores = Reduced Disease Activity
Time Frame: Day 29, Day 57, Day 85, Day 113, Day 141, Day 169
Population: Modified ITT Population
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
Scores on a scale
  Day 29: number analyzed (Participants) | 86 | 88
  Day 29 | -0.4 [-0.6 to -0.2] | -0.4 [-0.6 to -0.2]
  Day 57: number analyzed (Participants) | 84 | 90
  Day 57 | -0.6 [-0.8 to -0.4] | -0.7 [-0.9 to -0.4]
  Day 85: number analyzed (Participants) | 83 | 86
  Day 85 | -0.8 [-1.0 to -0.6] | -0.8 [-1.1 to -0.6]
  Day 113: number analyzed (Participants) | 81 | 85
  Day 113 | -0.8 [-1.0 to -0.5] | -1.0 [-1.2 to -0.7]
  Day 141: number analyzed (Participants) | 80 | 88
  Day 141 | -0.8 [-1.0 to -0.5] | -1.0 [-1.3 to -0.8]
  Day 169: number analyzed (Participants) | 79 | 85
  Day 169 | -0.9 [-1.1 to -0.6] | -1.1 [-1.4 to -0.9]

5. Secondary Outcome: Change From Baseline of DAS28-CRP: Tender Swollen Joint Count of at Least 3
Description: as for outcome 4
Time Frame: Day 29, Day 57, Day 85, Day 113, Day 141, Day 169
Population: Modified ITT Population with Baseline Tender plus Swollen Joint Count of at Least 3
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 57 | 63
Scores on a scale
  Day 29: number analyzed (Participants) | 52 | 58
  Day 29 | -0.5 [-0.8 to -0.2] | -0.6 [-0.9 to -0.3]
  Day 57: number analyzed (Participants) | 50 | 60
  Day 57 | -0.9 [-1.2 to -0.5] | -1.0 [-1.3 to -0.6]
  Day 85: number analyzed (Participants) | 50 | 57
  Day 85 | -1.1 [-1.5 to -0.7] | -1.2 [-1.5 to -0.8]
  Day 113: number analyzed (Participants) | 48 | 57
  Day 113 | -1.1 [-1.4 to -0.7] | -1.4 [-1.7 to -1.0]
  Day 141: number analyzed (Participants) | 48 | 59
  Day 141 | -1.2 [-1.5 to -0.8] | -1.5 [-1.8 to -1.1]
  Day 169: number analyzed (Participants) | 47 | 57
  Day 169 | -1.3 [-1.7 to -0.9] | -1.5 [-1.9 to -1.2]

6. Secondary Outcome: Change From Baseline of DAS28-CRP: Tender Swollen Joints Count Less Than 3
Description: as for outcome 4
Time Frame: Day 29, Day 57, Day 85, Day 113, Day 141, Day 169
Population: Modified ITT Population with Baseline Tender plus Swollen Joint Count of Less than 3
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 35 | 31
Scores on a scale
  Day 29: number analyzed (Participants) | 34 | 30
  Day 29 | -0.3 [-0.6 to 0.0] | -0.2 [-0.6 to 0.1]
  Day 57: number analyzed (Participants) | 34 | 30
  Day 57 | -0.2 [-0.5 to 0.1] | -0.2 [-0.5 to 0.1]
  Day 85: number analyzed (Participants) | 33 | 29
  Day 85 | -0.4 [-0.6 to -0.1] | -0.4 [-0.7 to -0.1]
  Day 113: number analyzed (Participants) | 33 | 28
  Day 113 | -0.3 [-0.6 to -0.0] | -0.3 [-0.6 to -0.1]
  Day 141: number analyzed (Participants) | 32 | 29
  Day 141 | -0.2 [-0.5 to 0.1] | -0.4 [-0.7 to -0.0]
  Day 169: number analyzed (Participants) | 32 | 28
  Day 169 | -0.3 [-0.5 to -0.0] | -0.5 [-0.7 to -0.2]

7. Secondary Outcome: Change From Baseline in the Joint Component of DAS28-CRP: In the Full Population
Description: The mean change from baseline at all measured time points up to Day 169 in the individual components of DAS28-CRP.
  Tender Joint: Count 1-28 Swollen Joint: Count 1-28
  Negative Scores = Reduced number of joints impacted Positive Scores = Increased number of joints impacted
Time Frame: Day 29, Day 57, Day 85, Day 113, Day 141, Day 169
Population: Modified intent to treat (ITT)
Measure: Mean (95% Confidence Interval); unit: Joint Count
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
Joint Count
  Day 29 - Tender Joint: number analyzed (Participants) | 90 | 90
  Day 29 - Tender Joint | -1.7 [-2.8 to -0.7] | -1.9 [-2.9 to -0.8]
  Day 29 - Swollen Joint: number analyzed (Participants) | 90 | 90
  Day 29 - Swollen Joint | -0.5 [-1.0 to 0.1] | -0.6 [-1.1 to -0.1]
  Day 57 - Tender Joint: number analyzed (Participants) | 87 | 92
  Day 57 - Tender Joint | -2.6 [-3.7 to -1.5] | -2.9 [-4.0 to -1.9]
  Day 57 - Swollen Joint: number analyzed (Participants) | 87 | 92
  Day 57 - Swollen Joint | -1.0 [-1.6 to -0.3] | -1.0 [-1.6 to -0.4]
  Day 85 - Tender Joint: number analyzed (Participants) | 85 | 89
  Day 85 - Tender Joint | -2.9 [-4.1 to -1.7] | -3.4 [-4.6 to -2.2]
  Day 85 - Swollen Joint: number analyzed (Participants) | 85 | 89
  Day 85 - Swollen Joint | -1.4 [-2.0 to -0.8] | -1.4 [-2.0 to -0.9]
  Day 113 - Tender Joint: number analyzed (Participants) | 83 | 87
  Day 113 - Tender Joint | -3.1 [-4.2 to -2.0] | -3.9 [-5.0 to -2.8]
  Day 113 - Swollen Joint: number analyzed (Participants) | 83 | 87
  Day 113 - Swollen Joint | -1.5 [-2.0 to -1.1] | -1.9 [-2.3 to -1.4]
  Day 141 - Tender Joint: number analyzed (Participants) | 82 | 89
  Day 141 - Tender Joint | -3.6 [-4.7 to -2.5] | -4.1 [-5.2 to -3.0]
  Day 141 - Swollen Joint: number analyzed (Participants) | 82 | 89
  Day 141 - Swollen Joint | -1.4 [-1.9 to -0.8] | -1.8 [-2.4 to -1.3]
  Day 169 - Tender Joint: number analyzed (Participants) | 81 | 87
  Day 169 - Tender Joint | -2.9 [-4.0 to -1.7] | -4.4 [-5.6 to -3.3]
  Day 169 - Swollen Joint: number analyzed (Participants) | 81 | 87
  Day 169 - Swollen Joint | -1.4 [-1.9 to -0.8] | -2.0 [-2.6 to -1.5]

8. Secondary Outcome: Change From Baseline in the CRP Component of DAS28-CRP: In the Full Population
Description: The mean change from baseline at all measured time points up to Day 169 in the individual components of DAS28-CRP.
  CRP: measured lab value
  Positive Number = Increased level of CRP Negative Number = Reduced Level of CRP
Time Frame: Day 29, Day 57, Day 85, Day 113, Day 141, Day 169
Population: Modified intent to treat (ITT)
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
mg/L
  Day 29 - CRP: number analyzed (Participants) | 87 | 90
  Day 29 - CRP | 0.3 [-1.4 to 2.0] | 0.6 [-1.0 to 2.3]
  Day 57 - CRP: number analyzed (Participants) | 85 | 91
  Day 57 - CRP | -0.1 [-2.1 to 1.8] | 1.8 [-0.1 to 3.6]
  Day 85 - CRP: number analyzed (Participants) | 83 | 88
  Day 85 - CRP | -0.2 [-5.0 to 4.5] | 3.0 [-1.6 to 7.6]
  Day 113 - CRP: number analyzed (Participants) | 81 | 86
  Day 113 - CRP | 1.6 [-0.8 to 4.1] | 0.3 [-2.1 to 2.6]
  Day 141 - CRP: number analyzed (Participants) | 80 | 89
  Day 141 - CRP | 3.5 [-1.7 to 8.8] | -0.2 [-5.2 to 4.7]
  Day 169 - CRP: number analyzed (Participants) | 79 | 86
  Day 169 - CRP | -0.2 [-1.8 to 1.3] | 0.0 [-1.5 to 1.5]

9. Secondary Outcome: Change From Baseline in the Assessment of Disease Activity Component of DAS28-CRP: In the Full Population
Description: The mean change from baseline at all measured time points up to Day 169 in the individual components of DAS28-CRP.
  Assesment of Disease Activity: 0-100 scale [100=Most severe]
  Positive Numbers = Increased Disease Activity Negative Numbers = Decreased Diseased activity
Time Frame: Day 29, Day 57, Day 85, Day 113, Day 141, Day 169
Population: Modified intent to treat (ITT)
Measure: Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
Scores on a Scale
  Day 29 - Assessment of Disease Activity: number analyzed (Participants) | 89 | 92
  Day 29 - Assessment of Disease Activity | -4.0 [-9.8 to 1.7] | -7.1 [-12.7 to -1.4]
  Day 57 - Assessment of Disease Activity: number analyzed (Participants) | 86 | 93
  Day 57 - Assessment of Disease Activity | -7.5 [-13.4 to -1.7] | -6.3 [-11.9 to -0.6]
  Day 85 - Assessment of Disease Activity: number analyzed (Participants) | 85 | 89
  Day 85 - Assessment of Disease Activity | -10.4 [-16.3 to -4.4] | -10.2 [-16.0 to -4.4]
  Day 113 - Assessment of Disease Activity: number analyzed (Participants) | 83 | 88
  Day 113 - Assessment of Disease Activity | -8.0 [-14.0 to -2.0] | -9.7 [-15.5 to -3.9]
  Day 141 - Assessment of Disease Activity: number analyzed (Participants) | 82 | 90
  Day 141 - Assessment of Disease Activity | -5.1 [-11.0 to 0.8] | -11.0 [-16.7 to -5.3]
  Day 169 - Assessment of Disease Activity: number analyzed (Participants) | 81 | 88
  Day 169 - Assessment of Disease Activity | -10.1 [-16.1 to -4.0] | -9.0 [-14.8 to -3.1]

10. Secondary Outcome: Change From Baseline in the Joint Component of DAS28-CRP: Tender Swollen Joints of at Least 3
Description: as for outcome 7
Time Frame: Day 29, Day 57, Day 85, Day 113, Day 141, Day 169
Population: Modified intent to treat (ITT) Population with Baseline Tender plus Swollen Joint Count of at least 3
Measure: Mean (95% Confidence Interval); unit: Joint Count
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 57 | 63
Joint Count
  Day 29 - Tender Joint: number analyzed (Participants) | 55 | 60
  Day 29 - Tender Joint | -2.8 [-4.5 to -1.0] | -3.0 [-4.7 to -1.3]
  Day 29 - Swollen Joint: number analyzed (Participants) | 55 | 60
  Day 29 - Swollen Joint | -0.7 [-1.5 to 0.2] | -0.9 [-1.7 to -0.1]
  Day 57 - Tender Joint: number analyzed (Participants) | 53 | 62
  Day 57 - Tender Joint | -4.1 [-5.9 to -2.3] | -4.8 [-6.5 to -3.0]
  Day 57 - Swollen Joint: number analyzed (Participants) | 53 | 62
  Day 57 - Swollen Joint | -1.5 [-2.6 to -0.5] | -1.6 [-2.6 to -0.5]
  Day 85 - Tender Joint: number analyzed (Participants) | 52 | 59
  Day 85 - Tender Joint | -4.4 [-6.3 to -2.4] | -5.4 [-7.2 to -3.6]
  Day 85 - Swollen Joint: number analyzed (Participants) | 52 | 59
  Day 85 - Swollen Joint | -2.1 [-3.1 to -1.1] | -2.2 [-3.2 to -1.3]
  Day 113 - Tender Joint: number analyzed (Participants) | 50 | 58
  Day 113 - Tender Joint | -4.8 [-6.6 to -2.9] | -6.0 [-7.7 to -4.2]
  Day 113 - Swollen Joint: number analyzed (Participants) | 50 | 58
  Day 113 - Swollen Joint | -2.3 [-3.2 to -1.5] | -2.9 [-3.7 to -2.2]
  Day 141 - Tender Joint: number analyzed (Participants) | 50 | 60
  Day 141 - Tender Joint | -5.7 [-7.5 to -3.8] | -6.4 [-8.2 to -4.7]
  Day 141 - Swollen Joint: number analyzed (Participants) | 50 | 60
  Day 141 - Swollen Joint | -2.2 [-3.1 to -1.3] | -3.0 [-3.8 to -2.1]
  Day 169 - Tender Joint: number analyzed (Participants) | 49 | 58
  Day 169 - Tender Joint | -4.6 [-6.5 to -2.7] | -6.7 [-8.5 to -4.9]
  Day 169 - Swollen Joint: number analyzed (Participants) | 49 | 58
  Day 169 - Swollen Joint | -2.2 [-3.1 to -1.3] | -3.1 [-4.0 to -2.3]

11. Secondary Outcome: Change From Baseline in the CRP Component of DAS28-CRP: Tender Swollen Joints of at Least 3
Description: as for outcome 8
Time Frame: Day 29, Day 57, Day 85, Day 113, Day 141, Day 169
Population: Modified intent to treat (ITT) Population with Baseline Tender plus Swollen Joint Count of at least 3
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 57 | 63
mg/L
  Day 29 - CRP: number analyzed (Participants) | 53 | 59
  Day 29 - CRP | -1.5 [-3.7 to 0.7] | -0.7 [-2.8 to 1.4]
  Day 57 - CRP: number analyzed (Participants) | 51 | 60
  Day 57 - CRP | -1.3 [-4.3 to 1.7] | 1.3 [-1.5 to 4.0]
  Day 85 - CRP: number analyzed (Participants) | 50 | 57
  Day 85 - CRP | -2.2 [-9.8 to 5.5] | 3.8 [-3.4 to 11.0]
  Day 113 - CRP: number analyzed (Participants) | 48 | 57
  Day 113 - CRP | 1.2 [-2.7 to 5.1] | -0.4 [-4.0 to 3.2]
  Day 141 - CRP: number analyzed (Participants) | 48 | 59
  Day 141 - CRP | 4.5 [-4.0 to 12.9] | -1.4 [-9.0 to 6.3]
  Day 169 - CRP: number analyzed (Participants) | 47 | 57
  Day 169 - CRP | -1.4 [-3.9 to 1.1] | -0.7 [-3.0 to 1.6]

12. Secondary Outcome: Change From Baseline in the Assessment of Disease Activity Component of DAS28-CRP: Tender Swollen Joints of at Least 3
Description: as for outcome 9
Time Frame: Day 29, Day 57, Day 85, Day 113, Day 141, Day 169
Population: Modified intent to treat (ITT) Population with Baseline Tender plus Swollen Joint Count of at least 3
Measure: Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 57 | 63
Score on a Scale
  Day 29 - Assessment of Disease Activity: number analyzed (Participants) | 54 | 61
  Day 29 - Assessment of Disease Activity | 0.6 [-6.9 to 8.1] | -3.5 [-10.7 to 3.7]
  Day 57 - Assessment of Disease Activity: number analyzed (Participants) | 52 | 62
  Day 57 - Assessment of Disease Activity | -3.5 [-11.5 to 4.5] | -6.5 [-14.0 to 1.1]
  Day 85 - Assessment of Disease Activity: number analyzed (Participants) | 52 | 59
  Day 85 - Assessment of Disease Activity | -7.5 [-15.5 to 0.4] | -7.7 [-15.3 to -0.1]
  Day 113 - Assessment of Disease Activity: number analyzed (Participants) | 50 | 58
  Day 113 - Assessment of Disease Activity | -6.6 [-14.4 to 1.3] | -9.1 [-16.5 to -1.6]
  Day 141 - Assessment of Disease Activity: number analyzed (Participants) | 50 | 60
  Day 141 - Assessment of Disease Activity | -1.2 [-9.0 to 6.7] | -8.1 [-15.5 to -0.7]
  Day 169 - Assessment of Disease Activity: number analyzed (Participants) | 49 | 58
  Day 169 - Assessment of Disease Activity | -6.7 [-14.9 to 1.5] | -7.8 [-15.5 to -0.0]

13. Secondary Outcome: Change From Baseline in the Joint Component of DAS28-CRP: Tender Swollen Joint Count Less Than 3
Description: as for outcome 7
Time Frame: Day 29, Day 57, Day 85, Day 113, Day 141, Day 169
Population: Modified intent to treat (ITT) Population with Baseline Tender plus Swollen Joint Count of Less than 3
Measure: Mean (95% Confidence Interval); unit: Joint Count
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 35 | 31
Joint Count
  Day 29 - Tender Joint: number analyzed (Participants) | 35 | 30
  Day 29 - Tender Joint | -0.1 [-0.9 to 0.6] | -0.2 [-0.9 to 0.6]
  Day 29 - Swollen Joint: number analyzed (Participants) | 35 | 30
  Day 29 - Swollen Joint | 0.1 [-0.2 to 0.3] | 0.1 [-0.2 to 0.4]
  Day 57 - Tender Joint: number analyzed (Participants) | 34 | 30
  Day 57 - Tender Joint | -0.2 [-0.9 to 0.6] | 0.1 [-0.6 to 0.9]
  Day 57 - Swollen Joint: number analyzed (Participants) | 34 | 30
  Day 57 - Swollen Joint | 0.2 [-0.1 to 0.4] | 0.0 [-0.2 to 0.3]
  Day 85 - Tender Joint: number analyzed (Participants) | 33 | 30
  Day 85 - Tender Joint | -0.5 [-1.3 to 0.2] | 0.1 [-0.7 to 0.8]
  Day 85 - Swollen Joint: number analyzed (Participants) | 33 | 30
  Day 85 - Swollen Joint | -0.0 [-0.3 to 0.2] | 0.1 [-0.2 to 0.4]
  Day 113 - Tender Joint: number analyzed (Participants) | 33 | 29
  Day 113 - Tender Joint | -0.4 [-1.2 to 0.3] | -0.5 [-1.3 to 0.3]
  Day 113 - Swollen Joint: number analyzed (Participants) | 33 | 29
  Day 113 - Swollen Joint | 0.0 [-0.3 to 0.3] | 0.1 [-0.2 to 0.4]
  Day 141 - Tender Joint: number analyzed (Participants) | 32 | 29
  Day 141 - Tender Joint | -0.2 [-1.0 to 0.6] | -0.2 [-1.0 to 0.6]
  Day 141 - Swollen Joint: number analyzed (Participants) | 32 | 29
  Day 141 - Swollen Joint | 0.2 [-0.1 to 0.5] | 0.3 [0.0 to 0.6]
  Day 169 - Tender Joint: number analyzed (Participants) | 32 | 29
  Day 169 - Tender Joint | -0.1 [-0.9 to 0.7] | -0.7 [-1.4 to 0.1]
  Day 169 - Swollen Joint: number analyzed (Participants) | 32 | 29
  Day 169 - Swollen Joint | 0.2 [-0.1 to 0.5] | -0.0 [-0.3 to 0.2]

14. Secondary Outcome: Change From Baseline in the CRP Component of DAS28-CRP: Tender Swollen Joint Count Less Than 3
Description: as for outcome 8
Time Frame: Day 29, Day 57, Day 85, Day 113, Day 141, Day 169
Population: Modified intent to treat (ITT) Population with Baseline Tender plus Swollen Joint Count of Less than 3
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 35 | 31
mg/L
  Day 29 - CRP: number analyzed (Participants) | 34 | 30
  Day 29 - CRP | 2.1 [-0.8 to 4.9] | 1.8 [-1.2 to 4.7]
  Day 57 - CRP: number analyzed (Participants) | 34 | 30
  Day 57 - CRP | 0.5 [-2.3 to 3.4] | 1.0 [-1.9 to 3.9]
  Day 85 - CRP: number analyzed (Participants) | 33 | 30
  Day 85 - CRP | 1.4 [-1.5 to 4.3] | 0.1 [-2.8 to 3.1]
  Day 113 - CRP: number analyzed (Participants) | 33 | 28
  Day 113 - CRP | 1.3 [-1.6 to 4.1] | 0.1 [-2.8 to 3.1]
  Day 141 - CRP: number analyzed (Participants) | 32 | 29
  Day 141 - CRP | 0.7 [-2.2 to 3.6] | 0.8 [-2.1 to 3.8]
  Day 169 - CRP: number analyzed (Participants) | 32 | 28
  Day 169 - CRP | 0.2 [-2.7 to 3.1] | 0.2 [-2.8 to 3.1]

15. Secondary Outcome: Change From Baseline in the Assessment of Disease Activity Component of DAS28-CRP: Tender Swollen Joint Count Less Than 3
Description: as for outcome 9
Time Frame: Day 29, Day 57, Day 85, Day 113, Day 141, Day 169
Population: Modified intent to treat (ITT) Population with Baseline Tender plus Swollen Joint Count of Less than 3
Measure: Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 35 | 31
Scores on a Scale
  Day 29 - Assessment of Disease Activity: number analyzed (Participants) | 35 | 30
  Day 29 - Assessment of Disease Activity | -10.3 [-19.3 to -1.4] | -11.8 [-21.3 to -2.3]
  Day 57 - Assessment of Disease Activity: number analyzed (Participants) | 34 | 30
  Day 57 - Assessment of Disease Activity | -12.4 [-21.4 to -3.4] | -4.8 [-14.3 to 4.7]
  Day 85 - Assessment of Disease Activity: number analyzed (Participants) | 33 | 29
  Day 85 - Assessment of Disease Activity | -14.0 [-23.0 to -5.0] | -13.5 [-23.0 to -4.0]
  Day 113 - Assessment of Disease Activity: number analyzed (Participants) | 33 | 29
  Day 113 - Assessment of Disease Activity | -9.1 [-18.1 to -0.0] | -11.1 [-20.6 to -1.5]
  Day 141 - Assessment of Disease Activity: number analyzed (Participants) | 32 | 29
  Day 141 - Assessment of Disease Activity | -10.6 [-19.8 to -1.5] | -15.3 [-24.8 to -5.7]
  Day 169 - Assessment of Disease Activity: number analyzed (Participants) | 32 | 29
  Day 169 - Assessment of Disease Activity | -13.8 [-23.0 to -4.6] | -10.9 [-20.5 to -1.4]

16. Secondary Outcome: Participants Who Achieve Minimally Clinically Important Change in ESSDAI in at Least 3 Points
Description: Proportion of participants who achieve a minimally clinically important change (of at least 3 points) in the ESSDAI at all measured time points up to Day 169.
Time Frame: Day 29, Day 57, Day 85, Day 113, Day 141, Day 169
Population: Modified intent to treat (ITT) Population
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
Percentage
  Day 29 | 37 [27.1 to 47.7] | 34.7 [25.3 to 45.2]
  Day 57 | 37 [27.1 to 47.7] | 44.2 [34.0 to 54.8]
  Day 85 | 48.9 [38.3 to 59.6] | 50.5 [40.1 to 60.9]
  Day 113 | 55.4 [44.7 to 65.8] | 50.5 [40.1 to 60.9]
  Day 141 | 51.1 [40.4 to 61.7] | 56.8 [46.3 to 67.0]
  Day 169 | 55.4 [44.7 to 65.8] | 57.9 [47.3 to 68.0]

17. Secondary Outcome: Participants Who Achieve Minimally Clinically Important Change in ESSDAI in at Least 5 Points
Description: Proportion of participants who achieve a minimally clinically important change (of at least 5 points) in the ESSDAI at all measured time points up to Day 169.
Time Frame: Day 29, Day 57, Day 85, Day 113, Day 141, Day 169
Population: Modified intent to treat (ITT) Population
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
Percentage
  Day 29 | 19.6 [12.0 to 29.1] | 13.7 [7.5 to 22.3]
  Day 57 | 26.1 [17.5 to 36.3] | 24.2 [16.0 to 34.1]
  Day 85 | 34.8 [25.1 to 45.4] | 32.6 [23.4 to 43.0]
  Day 113 | 37.0 [27.1 to 47.7] | 36.8 [27.2 to 47.4]
  Day 141 | 37.0 [27.1 to 47.7] | 36.8 [31.1 to 51.6]
  Day 169 | 35.9 [26.1 to 46.5] | 46.3 [36.0 to 56.8]

18. Secondary Outcome: Participants Who Achieve Minimally Clinically Important Change in ESSPRI in at Least 1 Point
Description: Proportion of participants who achieve a minimally clinically important change (of at least 1 point) in the ESSPRI at all measured time points up to Day 169.
Time Frame: Day 29, Day 57, Day 85, Day 113, Day 141, Day 169
Population: Modified intent to treat (ITT) Population
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
Percentage
  Day 29 | 31.5 [22.2 to 42.0] | 38.9 [29.1 to 49.5]
  Day 57 | 42.4 [32.1 to 53.1] | 47.4 [37.0 to 57.9]
  Day 85 | 44.6 [34.2 to 55.3] | 55.8 [45.2 to 66.0]
  Day 113 | 42.4 [32.1 to 53.1] | 52.6 [42.1 to 63.0]
  Day 141 | 40.2 [30.1 to 51.0] | 54.7 [44.2 to 65.0]
  Day 169 | 41.3 [31.1 to 52.1] | 52.6 [42.1 to 63.0]

19. Secondary Outcome: Change From Baseline at All Measured Time Points in the ESSDAI
Description: as for outcome 1
Time Frame: Day 29, Day 57, Day 85, Day 113, Day 141, Day 169
Population: Modified intent to treat (ITT) Population
Measure: Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
Percent Change from Baseline
  Day 29: number analyzed (Participants) | 89 | 92
  Day 29 | -10.9 [-22.3 to 0.54] | -12.6 [-23.71 to -1.39]
  Day 57: number analyzed (Participants) | 85 | 90
  Day 57 | -24.1 [-36.10 to -12.08] | -18.9 [-30.52 to -7.32]
  Day 85: number analyzed (Participants) | 85 | 90
  Day 85 | -26.0 [-38.81 to -13.17] | -25.4 [-37.76 to -13.01]
  Day 113: number analyzed (Participants) | 83 | 88
  Day 113 | -34.1 [-46.8 to -21.34] | -32.1 [-44.35 to -19.83]
  Day 141: number analyzed (Participants) | 82 | 89
  Day 141 | -29.7 [-43.02 to -16.31] | -37.0 [-49.81 to -24.12]
  Day 169: number analyzed (Participants) | 81 | 88
  Day 169 | -33.4 [-46.54 to -20.24] | -37.6 [-50.24 to -25.02]

20. Secondary Outcome: Change From Baseline at All Measured Time Points in the ESSPRI
Description: as for outcome 2
Time Frame: Day 29, Day 57, Day 85, Day 113, Day 141, Day 169
Population: Modified intent to treat (ITT) Population
Measure: Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
Score on a Scale
  Day 29: number analyzed (Participants) | 90 | 92
  Day 29 | -0.32 [-0.79 to 0.16] | -0.54 [-1.00 to -0.08]
  Day 57: number analyzed (Participants) | 87 | 93
  Day 57 | -0.81 [-1.32 to -0.31] | -0.82 [-1.31 to -0.33]
  Day 85: number analyzed (Participants) | 85 | 90
  Day 85 | -0.83 [-1.34 to -0.32] | -1.20 [-1.70 to -0.70]
  Day 113: number analyzed (Participants) | 83 | 88
  Day 113 | -0.79 [-1.32 to -0.26] | -1.37 [-1.88 to -0.86]
  Day 141: number analyzed (Participants) | 82 | 89
  Day 141 | -0.87 [-1.40 to -0.35] | -1.32 [-1.83 to -0.81]
  Day 169: number analyzed (Participants) | 81 | 88
  Day 169 | -1.03 [-1.55 to -0.50] | -1.30 [-1.80 to -0.79]

21. Secondary Outcome: Change From Baseline in Components of ESSDAI
Description: The EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) total score is calculated as the sum of scores for activity level for each domain.
  The EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) Scoring Algorithm.
  Domain: (Score for activity level) Constitutional: (No=0, Low=3, Moderate=6) Lymphadenopathy: (No=0, Low=4, Moderate=8, High=12) Glandular: (No=0, Low=2, Moderate=4) Articular: (No=0, Low=2, Moderate=4, High=6) Cutaneous: (No=0, Low=3, Moderate=6, High=9) Pulmonary: (No=0, Low=5, Moderate=10, High=15) Renal: (No=0, Low=5, Moderate=10, High=15) Muscular: (No=0, Low=6, Moderate=12, High=18) Peripheral Nervous System (PNS): (No=0, Low=5, Moderate=10, High=15) Central Nervous System (CNS): (No=0, Moderate=10, High=15) Haematological: (No=0, Low=2, Moderate=4, High=6) Biological: (No=0, Low=1, Moderate=2)
  (No = No Disease Activity, Low = Low Disease Activity, Moderate = Moderate Disease Activity, High = High Disease Activity)
Time Frame: Day 29, Day 57, Day 85, Day 113, Day 141 and Day 169
Population: Modified ITT Population
Measure: Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
Score on a Scale
  Day 29: Constitutional: number analyzed (Participants) | 89 | 92
  Day 29: Constitutional | -0.3 [-0.4 to -0.1] | -0.4 [-0.5 to -0.2]
  Day 29: Lymphadenopathy: number analyzed (Participants) | 89 | 92
  Day 29: Lymphadenopathy | -0.6 [-1.0 to -0.2] | -0.5 [-0.9 to -0.2]
  Day 29: Glandular: number analyzed (Participants) | 89 | 92
  Day 29: Glandular | -0.2 [-0.4 to 0.0] | -0.2 [-0.4 to 0.0]
  Day 29: Articular: number analyzed (Participants) | 89 | 91
  Day 29: Articular | -0.4 [-0.8 to 0.0] | -0.3 [-0.7 to 0.1]
  Day 29: Cutaneous: number analyzed (Participants) | 89 | 92
  Day 29: Cutaneous | -0.3 [-0.6 to -0.0] | -0.2 [-0.5 to 0.1]
  Day 29: Pulmonary: number analyzed (Participants) | 89 | 92
  Day 29: Pulmonary | 0.0 [-0.3 to 0.3] | 0.1 [-0.2 to 0.4]
  Day 29: Renal: number analyzed (Participants) | 89 | 92
  Day 29: Renal | -0.0 [-0.2 to 0.2] | -0.2 [-0.3 to 0.0]
  Day 29: Muscular: number analyzed (Participants) | 89 | 92
  Day 29: Muscular | -0.0 [-0.1 to 0.1] | -0.0 [-0.1 to 0.1]
  Day 29: Peripheral Nervous System: number analyzed (Participants) | 89 | 92
  Day 29: Peripheral Nervous System | -0.0 [-0.2 to 0.2] | 0.0 [-0.2 to 0.20]
  Day 29: Haematogical: number analyzed (Participants) | 89 | 92
  Day 29: Haematogical | 0.2 [-0.0 to 0.4] | 0.1 [-0.1 to 0.4]
  Day 29: Biological: number analyzed (Participants) | 89 | 92
  Day 29: Biological | 0.1 [-0.1 to 0.2] | 0.1 [-0.0 to 0.3]
  Day 57: Constitutional: number analyzed (Participants) | 85 | 90
  Day 57: Constitutional | -0.2 [-0.4 to -0.0] | -0.3 [-0.5 to -0.1]
  Day 57: Lymphadenopathy: number analyzed (Participants) | 85 | 90
  Day 57: Lymphadenopathy | -0.7 [-1.1 to -0.2] | -0.6 [-1.0 to -0.2]
  Day 57: Glandular: number analyzed (Participants) | 85 | 90
  Day 57: Glandular | -0.4 [-0.7 to -0.2] | -0.4 [-0.6 to -0.1]
  Day 57: Articular: number analyzed (Participants) | 85 | 90
  Day 57: Articular | -0.7 [-1.1 to -0.3] | -0.8 [-1.2 to -0.4]
  Day 57: Cutaneous: number analyzed (Participants) | 85 | 90
  Day 57: Cutaneous | -0.3 [-0.6 to -0.0] | -0.2 [-0.5 to 0.1]
  Day 57: Pulmonary: number analyzed (Participants) | 85 | 90
  Day 57: Pulmonary | -0.0 [-0.3 to 0.3] | 0.2 [-0.1 to 0.5]
  Day 57: Renal: number analyzed (Participants) | 85 | 90
  Day 57: Renal | -0.0 [-0.2 to 0.2] | -0.1 [-0.3 to 0.1]
  Day 57: Muscular: number analyzed (Participants) | 85 | 89
  Day 57: Muscular | -0.0 [-0.1 to 0.1] | -0.1 [-0.2 to -0.0]
  Day 57: Peripheral Nervous System: number analyzed (Participants) | 85 | 89
  Day 57: Peripheral Nervous System | -0.0 [-0.2 to 0.2] | 0.0 [-0.2 to 0.2]
  Day 57: Haematological: number analyzed (Participants) | 85 | 90
  Day 57: Haematological | 0.1 [-0.1 to 0.4] | 0.2 [-0.0 to 0.4]
  Day 57: Biological: number analyzed (Participants) | 81 | 84
  Day 57: Biological | -0.1 [-0.2 to 0.1] | 0.0 [-0.1 to 0.2]
  Day 85: Constitutional: number analyzed (Participants) | 85 | 90
  Day 85: Constitutional | -0.3 [-0.5 to -0.1] | -0.4 [-0.6 to -0.2]
  Day 85: Lymphadenopathy: number analyzed (Participants) | 85 | 90
  Day 85: Lymphadenopathy | -0.7 [-1.1 to -0.3] | -0.8 [-1.2 to -0.4]
  Day 85: Glandular: number analyzed (Participants) | 85 | 90
  Day 85: Glandular | -0.4 [-0.6 to -0.1] | -0.5 [-0.7 to -0.2]
  Day 85: Articular: number analyzed (Participants) | 85 | 90
  Day 85: Articular | -1.0 [-1.5 to -0.6] | -1.1 [-1.6 to -0.7]
  Day 85: Cutaneous: number analyzed (Participants) | 85 | 90
  Day 85: Cutaneous | -0.4 [-0.7 to -0.0] | -0.2 [-0.5 to 0.1]
  Day 85: Pulmonary: number analyzed (Participants) | 85 | 90
  Day 85: Pulmonary | 0.0 [-0.3 to 0.4] | 0.2 [-0.1 to 0.5]
  Day 85: Renal: number analyzed (Participants) | 85 | 90
  Day 85: Renal | -0.1 [-0.3 to 0.1] | -0.1 [-0.3 to 0.1]
  Day 85: Muscular: number analyzed (Participants) | 85 | 90
  Day 85: Muscular | -0.1 [-0.2 to 0.0] | -0.0 [-0.1 to 0.1]
  Day 85: Peripheral Nervous System: number analyzed (Participants) | 85 | 90
  Day 85: Peripheral Nervous System | -0.0 [-0.2 to 0.2] | 0.0 [-0.2 to 0.2]
  Day 85: Haematological: number analyzed (Participants) | 85 | 90
  Day 85: Haematological | 0.1 [-0.1 to 0.3] | 0.2 [-0.1 to 0.4]
  Day 85: Biological: number analyzed (Participants) | 85 | 90
  Day 85: Biological | 0.0 [-0.1 to 0.2] | 0.2 [0.0 to 0.3]
  Day 113: Constitutional: number analyzed (Participants) | 83 | 88
  Day 113: Constitutional | -0.3 [-0.5 to -0.0] | -0.3 [-0.5 to -0.1]
  Day 113: Lymphadenopathy: number analyzed (Participants) | 83 | 88
  Day 113: Lymphadenopathy | -0.8 [-1.2 to -0.4] | -0.9 [-1.3 to -0.5]
  Day 113: Glandular: number analyzed (Participants) | 83 | 88
  Day 113: Glandular | -0.5 [-0.7 to -0.3] | -0.5 [-0.8 to -0.3]
  Day 113: Articular: number analyzed (Participants) | 83 | 88
  Day 113: Articular | -1.3 [-1.8 to -0.8] | -1.3 [-1.7 to -0.8]
  Day 113: Cutaneous: number analyzed (Participants) | 83 | 88
  Day 113: Cutaneous | -0.4 [-0.7 to -0.1] | -0.4 [-0.7 to -0.1]
  Day 113: Pulmonary: number analyzed (Participants) | 83 | 88
  Day 113: Pulmonary | 0.0 [-0.3 to 0.4] | 0.1 [-0.2 to 0.5]
  Day 113: Renal: number analyzed (Participants) | 83 | 88
  Day 113: Renal | -0.1 [-0.3 to 0.1] | 0.0 [-0.2 to 0.2]
  Day 113: Muscular: number analyzed (Participants) | 83 | 88
  Day 113: Muscular | -0.0 [-0.1 to 0.1] | -0.1 [-0.2 to 0.0]
  Day 113: Peripheral Nervous System: number analyzed (Participants) | 83 | 88
  Day 113: Peripheral Nervous System | -0.0 [-0.2 to 0.2] | -0.0 [-0.2 to 0.1]
  Day 113: Haematological: number analyzed (Participants) | 83 | 88
  Day 113: Haematological | 0.1 [-0.2 to 0.3] | 0.2 [-0.0 to 0.4]
  Day 113: Biological: number analyzed (Participants) | 83 | 88
  Day 113: Biological | -0.0 [-0.2 to 0.1] | 0.1 [-0.0 to 0.3]
  Day 141: Constitutional: number analyzed (Participants) | 82 | 89
  Day 141: Constitutional | -0.2 [-0.4 to 0.0] | -0.4 [-0.6 to -0.2]
  Day 141: Lymphadenopathy: number analyzed (Participants) | 82 | 89
  Day 141: Lymphadenopathy | -0.6 [-1.1 to -0.2] | -0.9 [-1.4 to -0.5]
  Day 141: Glandular: number analyzed (Participants) | 82 | 89
  Day 141: Glandular | -0.5 [-0.7 to -0.2] | -0.6 [-0.8 to -0.4]
  Day 141: Articular: number analyzed (Participants) | 82 | 89
  Day 141: Articular | -1.2 [-1.7 to -0.8] | -1.4 [-1.9 to -1.0]
  Day 141: Cutaneous: number analyzed (Participants) | 82 | 89
  Day 141: Cutaneous | -0.4 [-0.7 to -0.1] | -0.5 [-0.8 to -0.3]
  Day 141: Pulmonary: number analyzed (Participants) | 82 | 89
  Day 141: Pulmonary | -0.0 [-0.4 to 0.3] | 0.1 [-0.2 to 0.4]
  Day 141: Renal: number analyzed (Participants) | 82 | 89
  Day 141: Renal | -0.0 [-0.2 to 0.2] | -0.1 [-0.3 to 0.1]
  Day 141: Muscular: number analyzed (Participants) | 82 | 89
  Day 141: Muscular | -0.1 [-0.2 to 0.0] | -0.1 [-0.2 to 0.0]
  Day 141: Peripheral Nervous System: number analyzed (Participants) | 82 | 89
  Day 141: Peripheral Nervous System | -0.1 [-0.3 to 0.1] | -0.0 [-0.2 to 0.1]
  Day 141: Haematological: number analyzed (Participants) | 82 | 89
  Day 141: Haematological | 0.1 [-0.1 to 0.4] | 0.1 [-0.1 to 0.4]
  Day 141: Biological: number analyzed (Participants) | 80 | 86
  Day 141: Biological | -0.0 [-0.2 to 0.1] | 0.1 [-0.0 to 0.2]
  Day 169: Constitutional: number analyzed (Participants) | 81 | 88
  Day 169: Constitutional | -0.3 [-0.5 to -0.1] | -0.4 [-0.6 to -0.2]
  Day 169: Lymphadenopathy: number analyzed (Participants) | 81 | 88
  Day 169: Lymphadenopathy | -0.9 [-1.3 to -0.5] | -1.1 [-1.4 to -0.7]
  Day 169: Glandular: number analyzed (Participants) | 81 | 88
  Day 169: Glandular | -0.4 [-0.6 to -0.1] | -0.5 [-0.8 to -0.3]
  Day 169: Articular: number analyzed (Participants) | 81 | 88
  Day 169: Articular | -1.4 [-1.8 to -0.9] | -1.8 [-2.2 to -1.4]
  Day 169: Cutaneous: number analyzed (Participants) | 81 | 88
  Day 169: Cutaneous | -0.3 [-0.7 to 0.0] | -0.5 [-0.9 to -0.2]
  Day 169: Pulmonary: number analyzed (Participants) | 81 | 88
  Day 169: Pulmonary | -0.0 [-0.4 to 0.3] | 0.1 [-0.2 to 0.4]
  Day 169: Renal: number analyzed (Participants) | 81 | 88
  Day 169: Renal | -0.0 [-0.2 to 0.2] | 0.0 [-0.2 to 0.2]
  Day 169: Muscular: number analyzed (Participants) | 81 | 88
  Day 169: Muscular | -0.0 [-0.1 to 0.1] | -0.1 [-0.2 to 0.0]
  Day 169: Peripheral Nervous: number analyzed (Participants) | 81 | 88
  Day 169: Peripheral Nervous | -0.1 [-0.3 to 0.1] | -0.0 [-0.2 to 0.2]
  Day 169: Haematological: number analyzed (Participants) | 81 | 88
  Day 169: Haematological | 0.1 [-0.2 to 0.3] | 0.3 [0.1 to 0.5]
  Day 169: Biological: number analyzed (Participants) | 81 | 88
  Day 169: Biological | 0.0 [-0.1 to 0.2] | 0.2 [0.0 to 0.3]

22. Secondary Outcome: Change From Baseline in ESSPRI Components
Description: as for outcome 2
Time Frame: Day 29, Day 57, Day 85, Day 113, Day 141, Day 169
Population: Modified ITT Population
Measure: Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
Score on a Scale
  Day 29: Dryness Score: number analyzed (Participants) | 90 | 92
  Day 29: Dryness Score | -0.21 [-0.76 to 0.34] | -0.26 [-0.80 to 0.28]
  Day 29: Fatigue Score: number analyzed (Participants) | 90 | 92
  Day 29: Fatigue Score | -0.57 [-1.18 to 0.03] | -1.01 [-1.60 to -0.42]
  Day 29: Pain Score: number analyzed (Participants) | 90 | 92
  Day 29: Pain Score | -0.34 [-0.96 to 0.27] | -0.53 [-1.13 to 0.07]
  Day 57: Dryness Score: number analyzed (Participants) | 87 | 93
  Day 57: Dryness Score | -0.92 [-1.51 to -0.33] | -0.52 [-1.09 to 0.05]
  Day 57: Fatigue Score: number analyzed (Participants) | 87 | 93
  Day 57: Fatigue Score | -1.09 [-1.70 to -0.48] | -1.22 [-1.81 to -0.63]
  Day 57: Pain Score: number analyzed (Participants) | 87 | 93
  Day 57: Pain Score | -0.60 [-1.24 to 0.05] | -0.90 [-1.52 to -0.27]
  Day 85: Dryness Score: number analyzed (Participants) | 85 | 90
  Day 85: Dryness Score | -0.68 [-1.25 to -0.11] | -0.91 [-1.46 to -0.36]
  Day 85: Fatigue Score: number analyzed (Participants) | 85 | 90
  Day 85: Fatigue Score | -1.27 [-1.91 to -0.63] | -1.56 [-2.18 to -0.94]
  Day 85: Pain Score: number analyzed (Participants) | 85 | 90
  Day 85: Pain Score | -0.70 [-1.35 to -0.05] | -1.31 [-1.93 to -0.68]
  Day 113: Dryness Score: number analyzed (Participants) | 83 | 88
  Day 113: Dryness Score | -0.74 [-1.36 to -0.12] | -1.19 [-1.79 to -0.60]
  Day 113: Fatigue Score: number analyzed (Participants) | 83 | 88
  Day 113: Fatigue Score | -1.02 [-1.65 to -0.39] | -1.76 [-2.37 to -1.15]
  Day 113: Pain Score: number analyzed (Participants) | 83 | 88
  Day 113: Pain Score | -0.76 [-1.40 to -0.11] | -1.37 [-1.99 to -0.74]
  Day 141: Dryness Score: number analyzed (Participants) | 82 | 89
  Day 141: Dryness Score | -0.89 [-1.49 to -0.28] | -1.05 [-1.63 to -0.46]
  Day 141: Fatigue Score: number analyzed (Participants) | 82 | 89
  Day 141: Fatigue Score | -1.18 [-1.83 to -0.53] | -1.73 [-2.36 to -1.11]
  Day 141: Pain Score: number analyzed (Participants) | 82 | 89
  Day 141: Pain Score | -0.70 [-1.34 to -0.07] | -1.39 [-2.00 to -0.78]
  Day 169: Dryness Score: number analyzed (Participants) | 81 | 88
  Day 169: Dryness Score | -0.84 [-1.46 to -0.23] | -1.04 [-1.63 to -0.44]
  Day 169: Fatigue Score: number analyzed (Participants) | 81 | 88
  Day 169: Fatigue Score | -1.28 [-1.93 to -0.64] | -1.57 [-2.19 to -0.95]
  Day 169: Pain Score: number analyzed (Participants) | 81 | 88
  Day 169: Pain Score | -1.11 [-1.75 to -0.47] | -1.45 [-2.06 to -0.83]

23. Secondary Outcome: Change From Baseline in Schirmer's Test
Description: The Mean change from baseline in Schirmer's Test at all measured time points up to day 169
  The length in millimeters that the strip wets during the 5 minute test period for each eye. Collection is done separately for each eye.
Time Frame: Day 85, Day 169
Population: Modified ITT Population
Measure: Mean (95% Confidence Interval); unit: millimeters
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
millimeters
  Day 85: Study Eye: number analyzed (Participants) | 81 | 85
  Day 85: Study Eye | 1.9 [-0.0 to 3.9] | 1.5 [-0.5 to 3.5]
  Day 85: Non-Study Eye: number analyzed (Participants) | 81 | 84
  Day 85: Non-Study Eye | 0.1 [-2.0 to 2.2] | 0.8 [-1.2 to 2.9]
  Day 85: Average of Both Eyes: number analyzed (Participants) | 81 | 84
  Day 85: Average of Both Eyes | 1.10 [-0.75 to 2.96] | 1.41 [-0.43 to 3.24]
  Day 169: Study Eye: number analyzed (Participants) | 73 | 75
  Day 169: Study Eye | 1.7 [-0.4 to 3.9] | 1.0 [-1.1 to 3.2]
  Day 169: Non-Study Eye: number analyzed (Participants) | 73 | 74
  Day 169: Non-Study Eye | 0.6 [-1.3 to 2.4] | 0.2 [-1.7 to 2.1]
  Day 169: Average of Both Eyes: number analyzed (Participants) | 73 | 74
  Day 169: Average of Both Eyes | 1.21 [-0.59 to 3.00] | 0.82 [-0.97 to 2.61]

24. Secondary Outcome: Change From Baseline in the Ocular Staining Score (OSS)
Description: The Mean change from baseline in OSS at all measured time points up to day 169
  Score of 0 = No Staining Score of 12 = diffuse staining
  The total score will be calculated as the sum of the score for these parameters for each eye.
  Medial Nasal Bulbar Conjunctiva (MNBC) [score scale: 0 - 3], Corneal (CORN) Staining of Punctate Epithelial Erosions (PEE) [score scale: 0 - 3], Lateral Temporal Bulbar Conjunctiva (LTBC) [score scale: 0 - 3], Patches of Confluent Staining (CONF) [score scale: 0 - 1], PEE observed in the pupil region, i.e. central 4mm diameter portion of the cornea (PUPL) [score scale: 0 - 1], one of more filaments seen anywhere on the cornea (FILA) [score scale: 0 - 1]
Time Frame: Day 85, Day 169
Population: Modified ITT Population
Measure: Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
Score on a Scale
  Day 85: Study Eye: number analyzed (Participants) | 81 | 86
  Day 85: Study Eye | -1.7 [-2.5 to -0.9] | -0.5 [-1.3 to 0.3]
  Day 85: Non-Study Eye: number analyzed (Participants) | 81 | 85
  Day 85: Non-Study Eye | -0.6 [-1.4 to 0.2] | 0.4 [-0.4 to 1.2]
  Day 85: Average of Both Eyes: number analyzed (Participants) | 81 | 85
  Day 85: Average of Both Eyes | -1.15 [-1.91 to -0.39] | -0.06 [-0.81 to 0.68]
  Day 169: Study Eye: number analyzed (Participants) | 73 | 75
  Day 169: Study Eye | -1.5 [-2.3 to -0.6] | -0.7 [-1.6 to 0.1]
  Day 169: Non-Study Eye: number analyzed (Participants) | 73 | 74
  Day 169: Non-Study Eye | -0.5 [-1.3 to 0.3] | 0.3 [-0.5 to 1.2]
  Day 169: Average of Both Eyes: number analyzed (Participants) | 73 | 74
  Day 169: Average of Both Eyes | -0.99 [-1.79 to -0.19] | -0.19 [-0.98 to 0.60]

25. Secondary Outcome: Change From Baseline in Tear Break-up Time
Description: The Mean change from baseline in Tear Break-up Time at all measured time points up to day 169
  The CRF collects the time in seconds to first appearance of a random dry spot on the corneal surface for 3 repetitions in each eye. The average time will calculated for each eye averaging the 3 measurements for each eye separately. In case only 2 measurements are available, the average of the 2 measurements will be calculated. In case there is only 1 measurement, that measurement will be used for the analysis.
Time Frame: Day 85, Day 169
Population: Modified ITT Population
Measure: Mean (95% Confidence Interval); unit: Seconds
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
Seconds
  Day 85: Study Eye: number analyzed (Participants) | 81 | 86
  Day 85: Study Eye | -0.13 [-0.99 to 0.73] | 0.18 [-0.67 to 1.04]
  Day 85: Non-Study Eye: number analyzed (Participants) | 81 | 86
  Day 85: Non-Study Eye | -0.70 [-1.59 to 0.18] | -0.12 [-1.01 to 0.76]
  Day 85: Average of Both Eyes: number analyzed (Participants) | 81 | 86
  Day 85: Average of Both Eyes | -0.41 [-1.24 to 0.43] | 0.09 [-0.74 to 0.92]
  Day 169: Study Eye: number analyzed (Participants) | 73 | 75
  Day 169: Study Eye | -0.23 [-1.11 to 0.64] | -0.32 [-1.19 to 0.56]
  Day 169: Non-Study Eye: number analyzed (Participants) | 73 | 74
  Day 169: Non-Study Eye | -0.79 [-1.62 to 0.03] | -0.62 [-1.46 to 0.21]
  Day 169: Average of Both Eyes: number analyzed (Participants) | 73 | 74
  Day 169: Average of Both Eyes | -0.50 [-1.32 to 0.31] | -0.43 [-1.25 to 0.39]

26. Secondary Outcome: Change From Baseline in Unstimulated Salivary Flow
Description: The mean change from baseline in unstimulated whole salivary flow at all measured time points up to Day 169.
Time Frame: Day 85, Day 169
Population: Modified ITT Population
Measure: Mean (95% Confidence Interval); unit: mL/min
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
mL/min
  Day 85: number analyzed (Participants) | 86 | 93
  Day 85 | 0.106 [-0.037 to 0.249] | 0.158 [0.022 to 0295]
  Day 169: number analyzed (Participants) | 81 | 87
  Day 169 | 0.051 [-0.100 to 0.203] | 0.105 [-0.042 to 0.251]

27. Secondary Outcome: Change From Baseline in Stimulated Salivary Flow
Description: The mean change from baseline in Stimulated whole salivary flow at all measured time points up to Day 169.
Time Frame: Day 85, Day 169
Population: Modified ITT Population
Measure: Mean (95% Confidence Interval); unit: mL/min
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 88 | 88
mL/min
  Day 85: number analyzed (Participants) | 82 | 87
  Day 85 | 0.11 [-0.039 to 0.262] | 0.169 [0.024 to 0.314]
  Day 169: number analyzed (Participants) | 77 | 81
  Day 169 | 0.056 [-0.104 to 0.216] | 0.108 [-0.048 to 0.263]

28. Secondary Outcome: Change From Baseline in Numeric Rating Scale for Mouth Dryness
Description: The mean change from baseline in participant symptoms using the Numeric Rating Scale (NRS) for mouth dryness at all measured time points up to Day 169.
  The oral and ocular dryness are each assessed by the patients with numeric rating scales from 0 to 10 with 0 representing no dryness and 10 representing maximal dryness
Time Frame: Day 1, 29, 57, 85, 113, 141, 169
Population: Modified ITT Population
Measure: Mean (Full Range); unit: Score on a Scale
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
Score on a Scale
  Day 29: number analyzed (Participants) | 89 | 92
  Day 29 | -0.8 [-8 to 3] | -0.5 [-7 to 6]
  Day 57: number analyzed (Participants) | 87 | 92
  Day 57 | -1.3 [-8 to 5] | -0.9 [-7 to 6]
  Day 85: number analyzed (Participants) | 85 | 90
  Day 85 | -1.3 [-9 to 4] | -1.1 [-6 to 8]
  Day 113: number analyzed (Participants) | 83 | 88
  Day 113 | -1.2 [-9 to 3] | -1.3 [-8 to 4]
  Day 141: number analyzed (Participants) | 82 | 90
  Day 141 | -1.3 [-8 to 5] | -1.1 [-6 to 6]
  Day 169: number analyzed (Participants) | 81 | 88
  Day 169 | -1.3 [-8 to 3] | -1.2 [-6 to 8]

29. Secondary Outcome: Change From Baseline in Numeric Rating Scale for Eye Dryness
Description: The mean change from baseline in patient symptoms using the Numeric Rating Scale (NRS) for eye dryness at all measured time points up to Day 169.
  The oral and ocular dryness are each assessed by the patients with numeric rating scales from 0 to 10 with 0 representing no dryness and 10 representing maximal dryness
Time Frame: Day 1, 29, 57, 85, 113, 141, 169
Population: Modified ITT Population
Measure: Mean (Full Range); unit: Score on a Scale
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
Score on a Scale
  Day 29: number analyzed (Participants) | 89 | 92
  Day 29 | -0.4 [-8 to 5] | -0.3 [-6 to 5]
  Day 57: number analyzed (Participants) | 87 | 92
  Day 57 | -0.9 [-7 to 5] | -0.6 [-6 to 5]
  Day 85: number analyzed (Participants) | 85 | 90
  Day 85 | -0.9 [-7 to 6] | -0.8 [-7 to 8]
  Day 113: number analyzed (Participants) | 83 | 88
  Day 113 | -1.0 [-7 to 7] | -1.1 [-8 to 4]
  Day 141: number analyzed (Participants) | 82 | 90
  Day 141 | -0.8 [-7 to 7] | -1.0 [-7 to 4]
  Day 169: number analyzed (Participants) | 81 | 88
  Day 169 | -0.9 [-5 to 6] | -1.0 [-7 to 5]

30. Secondary Outcome: Change From Baseline in Participant Assessment of Disease Activity
Description: The participant global assessment of disease activity are assessed with visual analog scales. The participant marks a vertical line through a horizontal line, where the beginning of the horizontal line represents the best situation, and the end of the horizontal line represents the very worst situation. The CRF collects the distance in millimeters from the start of the scale that is marked as well as the length of the scale in millimeters.
  In cases that the length of the scale is in less or more than 100 millimeters, then the participants measurement will be rescaled to the equivalent of 100 millimeters using the formula below:
  Rescale Measurement in mm = (measurement as reported on CRF in mm/length of the line on CRF in mm) * 100mm
  A negative score = participant assessment of disease activity has improved
  A positive score = participant assessment of disease activity has worsened
Time Frame: Day 29, 57, 85, 113, 141, 169
Population: Modified ITT Population
Measure: Mean (95% Confidence Interval); unit: Score on VAS 0-100mm scale
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
Score on VAS 0-100mm scale
  Day 29: number analyzed (Participants) | 89 | 92
  Day 29 | -4.0 [-9.8 to 1.7] | -7.1 [-12.7 to -1.4]
  Day 57: number analyzed (Participants) | 86 | 93
  Day 57 | -7.5 [-13.4 to -1.7] | -6.3 [-11.9 to -0.6]
  Day 85: number analyzed (Participants) | 85 | 89
  Day 85 | -10.4 [-16.3 to -4.4] | -10.2 [-16.0 to -4.4]
  Day 113: number analyzed (Participants) | 83 | 88
  Day 113 | -8.0 [-14.0 to -2.0] | -9.7 [-15.5 to -3.9]
  Day 141: number analyzed (Participants) | 82 | 90
  Day 141 | -5.1 [-11.0 to 0.8] | -11.0 [-16.7 to -5.3]
  Day 169: number analyzed (Participants) | 81 | 88
  Day 169 | -10.1 [-16.1 to -4.0] | -9.0 [-14.8 to -3.1]

31. Secondary Outcome: Change From Baseline in Physician Global Assessment of Disease Activity
Description: The physician global assessment of disease activity are assessed with visual analog scales. The physician marks a vertical line through a horizontal line, where the beginning of the horizontal line represents the best situation, and the end of the horizontal line represents the very worst situation. The CRF collects the distance in millimeters from the start of the scale that is marked as well as the length of the scale in millimeters.
  In cases that the length of the scale is in less or more than 100 millimeters, then the participants measurement will be rescaled to the equivalent of 100 millimeters using the formula below:
  Rescale Measurement in mm = (measurement as reported on CRF in mm/length of the line on CRF in mm) * 100mm
  A negative score = physician assessment of disease activity has improved
  A positive score = physician assessment of disease activity has worsened
Time Frame: Day 29, 57, 85, 113, 141, 169
Population: Modified ITT Population
Measure: Mean (95% Confidence Interval); unit: Score on VAS 0-100mm Scale
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
Score on VAS 0-100mm Scale
  Day 29: number analyzed (Participants) | 89 | 89
  Day 29 | -10.3 [-14.8 to -5.8] | -10.5 [-14.9 to -6.1]
  Day 57: number analyzed (Participants) | 86 | 92
  Day 57 | -16.2 [-20.8 to -11.7] | -16.7 [-21.1 to -12.3]
  Day 85: number analyzed (Participants) | 85 | 89
  Day 85 | -20.8 [-25.6 to -16.0] | -19.4 [-24.0 to -14.7]
  Day 113: number analyzed (Participants) | 82 | 87
  Day 113 | -22.8 [-27.9 to -17.8] | -19.8 [-24.6 to -14.9]
  Day 141: number analyzed (Participants) | 82 | 89
  Day 141 | -23.7 [-28.6 to -18.8] | -21.7 [-26.5 to -17.0]
  Day 169: number analyzed (Participants) | 81 | 87
  Day 169 | -23.0 [-27.8 to -18.2] | -23.7 [-28.3 to -19.0]

32. Secondary Outcome: Change From Baseline in Patient Fatigue
Description: The mean change from baseline in patient fatigue using Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue assessment of disease activity at all measured time points up to Day 169.
  PROMIS Fatigue instruments 10 Questions ranging from a score 0 to 40. Sum of the values gives you the raw sum. The raw is inputted into this formula to give you the raw score:
  Raw Score = (Raw sum*number of items on the short form)/(Number of items that were actually answered)
  Raw score is translated to a T-Score using a table. T-Score is used as the final score.
  The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. The standardized T-score is reported as the final score for each participant.
  A negative T Score = Better Prognosis A positive T Score = Worse prognosis
Time Frame: Day 29, 57, 85, 113, 141, 169
Population: Modified ITT Population
Measure: Mean (95% Confidence Interval); unit: T-Score
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
T-Score
  Day 29: number analyzed (Participants) | 90 | 92
  Day 29 | -3.08 [-5.22 to -0.95] | -3.99 [-6.09 to -1.88]
  Day 57: number analyzed (Participants) | 87 | 92
  Day 57 | -4.12 [-6.27 to -1.97] | -4.02 [-6.12 to -1.91]
  Day 85: number analyzed (Participants) | 85 | 90
  Day 85 | -4.85 [-7.05 to -2.64] | -5.48 [-7.64 to -3.32]
  Day 113: number analyzed (Participants) | 83 | 87
  Day 113 | -4.17 [-6.37 to -1.97] | -5.32 [-7.48 to -3.17]
  Day 141: number analyzed (Participants) | 82 | 89
  Day 141 | -4.84 [-7.06 to -2.62] | -5.68 [-7.85 to -3.52]
  Day 169: number analyzed (Participants) | 81 | 87
  Day 169 | -5.56 [-7.83 to -3.28] | -5.59 [-7.82 to -3.37]

33. Secondary Outcome: Change From Baseline in Female Sexual Function Using the Female Sexual Function Index (FSFI)
Description: For the FSFI, is a 19 item instrument used for assessing key dimensions of female sexual function over the past 4 weeks with 6 domains being analyzed. The specific domains (desire, arousal, lubrication, orgasm, satisfaction, and pain) analyzed in the FSFI are scored on a scale ranging from 0 to 5, with higher scores indicating better performance. Domain scores are calculated by summing the scores of the individual questions that make up the domain and multiplying the sum by the factor in the table below. The full scale score is the sum of the six domain scores.
  Full Scale Score range: 2.0(minimum score) - 36.0 (maximum score)
  Negative Score = Reduced functioning Positive Score = Improved functioning
Time Frame: Day 85, Day 169
Population: Modified ITT Population
Measure: Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 88 | 88
Scores on a Scale
  Day 85: number analyzed (Participants) | 62 | 58
  Day 85 | -2.44 [-5.67 to 0.78] | -1.56 [-4.90 to 1.77]
  Day 169: number analyzed (Participants) | 60 | 50
  Day 169 | -2.32 [-5.73 to 1.09] | -1.87 [-5.42 to 1.68]

34. Secondary Outcome: Change From Baseline in 36-item Short Form Health Survey (SF-36)
Description: The SF-36 determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health.
  Scores on each item are summed and averaged (range: 0=worst to 100=best). Increases from baseline indicate improvement
Time Frame: Day 85, Day 169
Population: Modified ITT Population
Measure: Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
Score on a Scale
  Day 85: Physical Function: number analyzed (Participants) | 89 | 92
  Day 85: Physical Function | 1.908 [-0.240 to 4.056] | 1.523 [-0.568 to 3.614]
  Day 85: Role Physical: number analyzed (Participants) | 90 | 92
  Day 85: Role Physical | 5.248 [3.112 to 7.383] | 4.416 [2.321 to 6.511]
  Day 85: Bodily Pain: number analyzed (Participants) | 90 | 92
  Day 85: Bodily Pain | 3.200 [0.910 to 5.490] | 3.721 [1.464 to 5.978]
  Day 85: General Health: number analyzed (Participants) | 90 | 92
  Day 85: General Health | 4.042 [1.938 to 6.146] | 3.409 [1.363 to 5.456]
  Day 85: Vitality: number analyzed (Participants) | 90 | 92
  Day 85: Vitality | 3.827 [1.269 to 6.384] | 3.859 [1.335 to 6.382]
  Day 85: Social Functioning: number analyzed (Participants) | 90 | 92
  Day 85: Social Functioning | 3.020 [0.296 to 5.744] | 4.771 [2.117 to 7.426]
  Day 85: Role-Emotional: number analyzed (Participants) | 90 | 92
  Day 85: Role-Emotional | 3.024 [0.214 to 5.834] | 4.834 [2.093 to 7.576]
  Day 85: Mental Health: number analyzed (Participants) | 90 | 92
  Day 85: Mental Health | 2.942 [0.458 to 5.425] | 2.287 [-0.135 to 4.709]
  Day 85: Physical component Summary: number analyzed (Participants) | 89 | 92
  Day 85: Physical component Summary | 3.430 [1.615 to 5.244] | 2.686 [0.904 to 4.468]
  Day 85: Mental component Summary: number analyzed (Participants) | 89 | 92
  Day 85: Mental component Summary | 2.693 [0.160 to 5.226] | 3.672 [1.208 to 6.136]
  Day 169: Physical Function: number analyzed (Participants) | 82 | 91
  Day 169: Physical Function | 2.927 [0.593 to 5.261] | 1.742 [-0.505 to 3.989]
  Day 169: Role-Physical: number analyzed (Participants) | 83 | 91
  Day 169: Role-Physical | 5.853 [3.756 to 7.949] | 4.626 [2.604 to 6.649]
  Day 169: Bodily Pain: number analyzed (Participants) | 83 | 91
  Day 169: Bodily Pain | 3.842 [1.432 to 6.252] | 3.458 [1.114 to 5.801]
  Day 169: General Health: number analyzed (Participants) | 83 | 91
  Day 169: General Health | 3.880 [1.700 to 6.060] | 3.764 [1.665 to 5.862]
  Day 169: Vitality: number analyzed (Participants) | 82 | 91
  Day 169: Vitality | 3.742 [1.160 to 6.324] | 4.523 [2.005 to 7.041]
  Day 169: Social functioning: number analyzed (Participants) | 83 | 91
  Day 169: Social functioning | 4.125 [1.320 to 6.929] | 4.471 [1.773 to 7.169]
  Day 169: Role-Emotional: number analyzed (Participants) | 83 | 91
  Day 169: Role-Emotional | 4.653 [1.943 to 7.364] | 4.930 [2.334 to 7.526]
  Day 169: Mental Health: number analyzed (Participants) | 83 | 91
  Day 169: Mental Health | 2.375 [-0.116 to 4.866] | 2.972 [0.581 to 5.363]
  Day 169: Physical Component Summary: number analyzed (Participants) | 81 | 91
  Day 169: Physical Component Summary | 3.998 [2.045 to 5.951] | 2.650 [0.756 to 4.543]
  Day 169: Mental Component Summary: number analyzed (Participants) | 81 | 91
  Day 169: Mental Component Summary | 2.940 [0.368 to 5.512] | 4.112 [1.648 to 6.577]

35. Secondary Outcome: Geometric Mean of Trough Concentration (Cmin) of Abatacept
Description: Geometric mean of trough concentration (Cmin) of abatacept at all measured time points.
Time Frame: Day 29, 85, 113, 141, 169
Population: Pharmacokinetic (PK) Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 0
µg/mL
  Day 29: number analyzed (Participants) | 68 | 0
  Day 29 | 21.401 (36) |
  Day 85: number analyzed (Participants) | 72 | 0
  Day 85 | 27.543 (38.4) |
  Day 113: number analyzed (Participants) | 72 | 0
  Day 113 | 25.567 (42.1) |
  Day 141: number analyzed (Participants) | 74 | 0
  Day 141 | 25.870 (40.8) |
  Day 169: number analyzed (Participants) | 74 | 0
  Day 169 | 24.522 (42.7) |

36. Secondary Outcome: Percentage of Participants With a Positive Antibody Response
Description: Percentage of participants with at least one positive immunogenicity response up to Day 169 and during 3 months follow up (for participants who discontinue during the 6-months double-blind).
Time Frame: Day 85 db, day 169 db, post treatment day 85
Population: Immunogenicity Analysis Population
Measure: Number; unit: Percentage
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 90 | 43
Percentage
  Study Day 169: number analyzed (Participants) | 81 | 0
  Study Day 169 | 1.2 |
  Post Treatment Day 85 (DB): number analyzed (Participants) | 5 | 0
  Post Treatment Day 85 (DB) | 0 |
  Post Treatment Day 169 (DB): number analyzed (Participants) | 4 | 0
  Post Treatment Day 169 (DB) | 0 |

37. Secondary Outcome: Summary of Adverse Events: Double Blind Period
Description: Percentage of participants with adverse events, deaths, serious adverse events and adverse events leading to discontinuation
Time Frame: Day 1 up to first dose of Open Label Treatment Period (OLTP) abatacept or up to 56 post last dose in double -blind for those not in OL.
Population: As-Treated Population
Measure: Number; unit: Percentage
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 92 | 95
Percentage
  Adverse Events (AEs) | 85.9 | 71.6
  Deaths | 0 | 1.1
  Serious Adverse Events | 9.8 | 3.2
  Discontinuation due to AEs | 3.3 | 2.1

38. Secondary Outcome: Laboratory Marked Abnormalities: Double Blind Period
Description: Laboratory values meeting the marked abnormality criteria
Time Frame: Day 1 up to first dose of OL abatacept or up to 56 post last dose in double -blind for those not in OL.
Population: As-Treated Analysis Population
Measure: Number; unit: Percentage
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period
Number analyzed (Participants) | 91 | 95
Percentage
  Hematocrit High | NA — Not Evaluated | NA — Not Evaluated
  Hematocrit Low | 0 | 0
  Hemoglobin High | NA — Not Evaluated | NA — Not Evaluated
  Hemoglobin Low | 0 | 0
  Platelet count High | 0 | 0
  Platelet count low | 0 | 0
  Leukocytes high | 1.1 | 0
  Leukocytes low | 12.1 | 8.4
  Basophils high | 0 | 0
  Basophils Low | NA — Not Evaluated | NA — Not Evaluated
  Eosinophils High | 4.4 | 1.1
  Eosinophils Low | NA — Not Evaluated | NA — Not Evaluated
  lymphocytes high | 0 | 0
  lymphocytes low | 9.9 | 14.7
  Monocytes high | 0 | 0
  Monocytes Low | NA — Not Evaluated | NA — Not Evaluated
  Neutrophils+Bands High | NA — Not Evaluated | NA — Not Evaluated
  Neutrophils+Bands Low | 6.6 | 1.1
  Alanine Aminotransferase High | 1.1 | 2.1
  Alkaline Phosphatase HIgh | 0 | 0
  Aspartate Aminotransferase High | 1.1 | 3.2
  Bilirubin, Total High | 0 | 0
  G-Glutamyl Transferase High | 6.6 | 1.1
  Blood Urea Nitrogen High | 1.1 | 1.1
  Creatinine High | 0 | 0
  Calcium High | 0 | 0
  Calcium Low | 1.1 | 0
  Chloride High | 0 | 0
  Chloride Low | 1.1 | 0
  Phosphorus High | 0 | 0
  Phosphorus Low | 0 | 1.1
  Potassium High | 0 | 0
  Potassium Low | 1.1 | 0
  Sodium High | 0 | 1.1
  Sodium Low | 2.2 | 0
  Glucose, Serum High | 0 | 1.1
  Glucose, Serum Low | 2.2 | 5.3
  Albumin High | NA — Not Evaluated | NA — Not Evaluated
  Albumin Low | 2.2 | 1.1
  Protein, Total High | 2.2 | 3.2
  Protein, Total Low | 1.1 | 0
  Creatine Kinase High | 0 | 4.2
  Blood, Urine High | 14.3 | 9.5
  Blood, Urine Low | NA — Not Evaluated | NA — Not Evaluated
  Glucose, Urine High | 0 | 0
  Glucose, Urine Low | NA — Not Evaluated | NA — Not Evaluated
  Protein, Urine High | 2.2 | 3.2

39. Secondary Outcome: Percentage of Participants With a Positive Antibody Response in the Cumulative Abatacept Period
Description: Percentage of participants with at least one positive immunogenicity response On Day 365 (end of Open label treatment period) and day 85 post open label follow up period.
Time Frame: Day 365, post open label treatment day 85
Population: Immunogenicity Analysis Population
Measure: Number; unit: Percentage
Groups:
- Abatacept - Cumulative Open Label Treatment Period: Cumulative Open Label Treatment Period SC injection 125mg/mL in 1 mL pre-filled syringe
Arm/Group | Abatacept - Cumulative Open Label Treatment Period
Number analyzed (Participants) | 177
Percentage
  Study Day 365: number analyzed (Participants) | 142
  Study Day 365 | 2.1
  Post Treatment Day 85 (OL): number analyzed (Participants) | 125
  Post Treatment Day 85 (OL) | 43.2

40. Secondary Outcome: Summary of Adverse Events: Cumulative Abatacept Period
Description: as for outcome 37
Time Frame: Day 365 and 3 months of follow up approximately 450 Days
Population: Cumulative Abatacept Population
Measure: Number; unit: Percentage
Groups:
- Cumulative Treatment Period: Cumulative Open Label Treatment Period SC injection 125mg/mL in 1 mL pre-filled syringe
Arm/Group | Cumulative Treatment Period
Number analyzed (Participants) | 178
Percentage
  Adverse Events (AEs) | 78.7
  Deaths | 0.6
  Serious Adverse Events (SAEs) | 14.6
  Discontinuation due to AEs | 5.6
  Related Serious Adverse Events | 3.4
  Discontinued due to SAEs | 3.4
  Related AEs | 40.4

41. Secondary Outcome: Laboratory Marked Abnormalities: Cumulative Abatacept Period
Description: Laboratory values meeting the marked abnormality criteria
Time Frame: Day 365 and 3 months of follow up approximately 450 Days
Population: Cumulative Abatacept Population
Measure: Number; unit: Percentage
Groups:
- Cumulative Open Label Treatment Period: Cumulative Open Label Treatment Period SC injection 125mg/mL in 1 mL pre-filled syringe
Arm/Group | Cumulative Open Label Treatment Period
Number analyzed (Participants) | 177
Percentage
  Hematocrit High | NA — Not Evaluated
  Hematocrit Low | 0
  Hemoglobin High | NA — Not Evaluated
  Hemoglobin Low | 0.6
  Platelet count High | 0
  Platelet count low | 0.6
  Leukocytes high | 0.6
  Leukocytes low | 18.6
  Basophils high | 0.6
  Basophils Low | NA — Not Evaluated
  Eosinophils High | 5.6
  Eosinophils Low | NA — Not Evaluated
  lymphocytes high | 0
  lymphocytes low | 12.4
  Monocytes high | 0
  Monocytes Low | NA — Not Evaluated
  Neutrophils+Bands High | NA — Not Evaluated
  Neutrophils+Bands Low | 7.3
  Alanine Aminotransferase High | 1.7
  Alkaline Phosphatase HIgh | 0.6
  Aspartate Aminotransferase High | 1.1
  Bilirubin, Total High | 0
  G-Glutamyl Transferase High | 5.6
  Blood Urea Nitrogen High | 1.7
  Creatinine High | 0.6
  Calcium High | 0
  Calcium Low | 1.1
  Chloride High | 0
  Chloride Low | 1.1
  Phosphorus High | 0.6
  Phosphorus Low | 1.1
  Potassium High | 0.6
  Potassium Low | 0.6
  Sodium High | 0.6
  Sodium Low | 1.7
  Glucose, Serum High | 0.6
  Glucose, Serum Low | 5.1
  Albumin High | NA — Not Evaluated
  Albumin Low | 1.7
  Protein, Total High | 4.0
  Protein, Total Low | 0.6
  Creatine Kinase High | 2.3
  Blood, Urine High | 14.7
  Blood, Urine Low | NA — Not Evaluated
  Glucose, Urine High | 0
  Glucose, Urine Low | NA — Not Evaluated
  Protein, Urine High | 5.6
  WBC, Urine High: number analyzed (Participants) | 1
  WBC, Urine High | 100.0

ADVERSE EVENTS:
Time Frame: First dose to 169 days past open label period
Groups:
- Abatacept - Open Label Treatment Period: Open Label Treatment Period SC injection 125mg/mL in 1 mL pre-filled syringe
Arm/Group | Abatacept - Double Blind Treatment Period | Placebo - Double Blind Treatment Period | Abatacept - Open Label Treatment Period
All-Cause Mortality (participants affected / at risk) | 0/92 | 1/95 | 1/178
Serious Adverse Events (participants affected / at risk) | 9/92 | 3/95 | 19/178
Other Adverse Events (participants affected / at risk) | 47/92 | 40/95 | 61/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Abatacept - Double Blind Treatment Period (N=92) | Placebo - Double Blind Treatment Period (N=95) | Abatacept - Open Label Treatment Period (N=178)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0/165
Angina pectoris (Cardiac disorders) | 0 | 0 | 1/165
Pericarditis (Cardiac disorders) | 0 | 0 | 1/165
Prinzmetal angina (Cardiac disorders) | 1 | 0 | 0/165
Colitis (Gastrointestinal disorders) | 0 | 1 | 0/165
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0/165
Pyrexia (General disorders) | 0 | 0 | 1/165
Sudden cardiac death (General disorders) | 0 | 0 | 1/165
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1/165
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1/165
Hepatic cyst ruptured (Hepatobiliary disorders) | 1 | 0 | 0/165
Anaphylactoid reaction (Immune system disorders) | 1 | 0 | 0/165
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0/165
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 1/165
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 1/165
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0/165
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1/165
Septic shock (Infections and infestations) | 0 | 1 | 0/165
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1/165
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0/165
Hip deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1/165
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0/165
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1/165
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1/165
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1/165
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1/165
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0/165
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1/165
Facial paralysis (Nervous system disorders) | 0 | 0 | 1/165
Migraine (Nervous system disorders) | 0 | 0 | 1/165
Syncope (Nervous system disorders) | 0 | 0 | 1/165
Device dislocation (Product Issues) | 0 | 0 | 2/165
Depression (Psychiatric disorders) | 0 | 0 | 1/165
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1/165
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept - Double Blind Treatment Period (N=92) | Placebo - Double Blind Treatment Period (N=95) | Abatacept - Open Label Treatment Period (N=165)
Abdominal pain upper (Gastrointestinal disorders) | 5 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 11 | 4 | 9
Nausea (Gastrointestinal disorders) | 9 | 4 | 1
Nasopharyngitis (Infections and infestations) | 11 | 18 | 22
Upper respiratory tract infection (Infections and infestations) | 9 | 7 | 15
Urinary tract infection (Infections and infestations) | 6 | 8 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 2 | 4
Headache (Nervous system disorders) | 10 | 9 | 9
Insomnia (Psychiatric disorders) | 5 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT02915159/SAP_000.pdf
  • Study Protocol (2016-08-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT02915159/Prot_001.pdf